CLINICAL TRIAL: NCT06559956
Title: Non-inferiority Analysis of Daytime Versus Overnight Polysomnography for Hypoglossal Nerve Stimulation Titration in Obstructive Sleep Apnea
Brief Title: Non-inferiority Analysis of Two Titration Methods for Hypoglossal Nerve Stimulation Therapy
Acronym: DOT-PSG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: B3002024000122
Record Dates: First submitted 2024-07-29; First posted 2024-08-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Apnea
Keywords: hypoglossal nerve stimulation; titration polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Overnight titration polysomnography cohort: A cohort of OSA patients treated with HNS that previously underwent an overnight titration PSG as part of the routine clinical care pathway
- Daytime titration polysomnography cohort: OSA patients treated with HNS that recently underwent or will be undergoing the newly introduced titration method, which is a daytime titration PSG.
  Interventions: Other: Daytime titration polysomnography

INTERVENTIONS:
Other: Daytime titration polysomnography — A titration polysomnography assesses the device settings and, if necessary, the stimulation strength will be adjusted based on observed respiratory events and/or snoring. Patients in the daytime titration PSG cohort were instructed to refrain from sleeping during the night, and in the morning, they were permitted to sleep in a soundproof room without daylight at the sleep lab.
  Groups: Daytime titration polysomnography cohort

SUMMARY:
Hypoglossal nerve stimulation (HNS) therapy (Inspire system) is intended for the treatment of patients with moderate to severe obstructive sleep apnea (OSA) who cannot be effectively treated with the first-line treatment options.

Approximately 3 months after activation of HNS therapy, a fine-tuning sleep study is performed. To date, the standard of care involves an in-laboratory overnight titration PSG, which assesses the device settings and, if necessary, the stimulation strength will be adjusted based on observed respiratory events and/or snoring. Considering the growing patient population, the performance of these overnight titrations can become logistically challenging and labor-intensive. Recently, the feasibility of using a daytime PSG as an alternative to a conventional overnight PSG for titration of HNS therapy was demonstrated.

The aim of this study is to further investigate this technique by performing a non-inferiority analysis of daytime versus overnight PSG for titration of HNS therapy in patients with OSA.

DETAILED DESCRIPTION:
This study is a prospective and retrospective, single-center non-inferiority study. The study population consists of two cohorts: (1) OSA patients treated with HNS that previously underwent an overnight titration PSG as part of the routine clinical care pathway and (2) OSA patients treated with HNS that recently underwent or will be undergoing a daytime titration PSG.

Data collection will include polysomnographic data, home sleep test data, therapy usage, device data and questionnaires (Epworth Sleepiness Scale, Functional Outcomes of Sleep Questionnaire-30, Visual Analogue Scale (VAS) snoring. Data will be collected from different visits including: pre-implant, implant, activation, titration, follow-up (6 and 12 months post-implantation).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OSA and implanted with HNS therapy (Inspire system)
* Cohort 1: Patients that previously underwent an overnight titration PSG as part of their routine clinical care at the Antwerp University Hospital
* Cohort 2: Patients that recently underwent or will be undergoing a daytime titration PSG at the Antwerp University Hospital
* Able to give informed consent

Exclusion Criteria:

* Not able to understand the language of the questionnaires

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with OSA and implanted with HNS therapy (Inspire system)
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the delta apnea-hypopnea index (AHI) between the two cohorts as measured by a titration polysomnography | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  The AHI is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow) per hour of sleep

SECONDARY OUTCOMES:
Percent of patients that reach treatment success defined by a 50% reduction in AHI and an on therapy AHI of < 20 events/h OR an on therapy AHI of < 15 events/h | At the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  AHI is determined during a polysomnography
Treatment AHI as measured during a titration polysomnography | At the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  The treatment AHI, also called the titrated AHI, is the AHI measurement from the portion of sleep when therapy is under therapeutic setting found for home use
Full-night AHI as measured during a titration polysomnography | At the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  Full-night AHI is the AHI determined from the complete titration polysomnography.
Percent of time spent in each sleep stage as measured during a titration polysomnography | At the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  Sleep architecture is the structure of the sleeping pattern, including rapid-eye movement sleep (REM) and nonREM sleep, and is measured during a polysomnography
Percent of time spent in different body positions during a titration polysomnography | At the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  The body position is recorded during a polysomnography
Delta oxygen desaturation index (ODI) as measured by a polysomnography | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  The ODI represents the average number of desaturation episodes (≥3%) per hour sleep and will be determined during a polysomnography
Daytime sleepiness measured by the Epworth Sleepiness Scale (ESS) questionnaire | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  The ESS questionnaire assesses the probability of falling asleep in various settings and situations in daily life. This questionnaire consists of eight questions which can be scored on a four-point Likert-type scale. The lowest score (zero) suggests that the described incident is absent and the highest score (three) suggests the presence of this event. The summation of the eight items can range from 0 to 24.
Disease-specific quality of life as measured by the Functional Outcomes of Sleep Questionnaire-30 (FOSQ-30) questionnaire | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  The FOSQ-30 is a disease-specific quality of life questionnaire that determines functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment. The total score equals the mean scores for each subscale (5 in total) multiplied by the number of subscales answered (total score range 5-20, with higher scores indicating better functional status
Degree of snoring measured by the Visual Analogue Scale (VAS) questionnaire | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  Snoring intensity is evaluated using a 10 cm visual analogue scale (VAS) from 0 to 10: 0 represents no snoring, 1-3 represents minimally annoying, 4-6 represents moderately annoying, 7-9 represents annoying, and 10 represents extremely annoying
Therapy adherence defined by the amount of hours therapy usage per night | At the postoperative titration follow-up (approximately 3 months after activation of the therapy) and 12 months follow-up
  Average hours of therapy use per night can be retrieved from data stored in the device
Delta sleep apnea specific hypoxic burden (SASHB) derived from a titration polysomnography | From baseline to the postoperative titration follow-up (approximately 3 months after activation of the therapy)
  SASHB is calculated as the oxygen desaturation "area under the curve" in association with individual apneas and hypopneas

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No